CLINICAL TRIAL: NCT04775303
Title: An Investigator Initiated Multi-center Phase 4 Clinical Trial to Evaluate the Clinical Efficacy of Cyclosporine 0.1% (Ikervis®) for Moderate to Severe Dry Eye Patients With Inadequate Effects From Previous Treatment (IKE-03, Switching Study)
Brief Title: A Clinical Trial to Evaluate the Clinical Efficacy of Cyclosporine 0.1% (Ikervis®) for Moderate to Severe Dry Eye Patients. (IKE-03-SWITCHING)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-1156
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Moderate to Severe Dry Eye
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Cyclosporine 0.1% (Ikervis®) eye drop - one drop once daily
  Interventions: Drug: Cyclosporine 0.1% (Ikervis®) eye drop

INTERVENTIONS:
Drug: Cyclosporine 0.1% (Ikervis®) eye drop — One drop of Cyclosporine 0.1% (Ikervis®) eye drop once daily for 12 weeks

SUMMARY:
A clinical trial to evaluate the efficacy and safety of Cyclosporine 0.1% (Ikervis®) for moderate to severe dry eye patients who changed to Cyclosporine 0.1% eye drop(Ikervis®) due to lack of treatment effects of the previous Cyclosporine 0.05% eye drop.

DETAILED DESCRIPTION:
Eligible patients who agree to participate in the clinical trial in writing will be administered Cyclosporine 0.1% eye drop(Ikervis®) one drop once daily for 12 weeks. Efficacy and safety will be evaluated at baseline, 4 weeks, 8 weeks, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 19 and less than 80 years old
2. A patient with moderate or severe dry eye who has used Cyclosporine 0.05% eye drop for more than 3 months and has no or insufficient treatment effect

   - No or insufficient treatment effect should meet the following criteria through tests used to diagnose dry eyes
   * A SANDE (Symptom Assessment in Dry Eye) score of 40 or more on the severity and frequency of dry eye symptoms.
   * Cornea staining score (NEI scale) 3 or more points
   * Tear Break Up Time(TBUT) 10 seconds or less
   * Tear volume tested by Tear Meniscometry less than 5mm
   * Has One or more of the dry eye symptoms; stinging, irritating, itching or blurred vision.
   * Use of diquafosol tetrasodium 3% eye drop and/or artificial tears are allowed with no change of products and dosage throughout the trial period
3. A person who voluntarily agrees in writing to participate in this clinical trial

Exclusion Criteria:

1. Use of eye drops within four weeks of the consent date such as steroids, glaucoma, allergies and anti-inflammatory drugs, etc.
2. Systematic steroid within four weeks of the consent date
3. Patients with pterygium
4. Start new immunosuppressive drugs or change in dosage that can affect immune function within four weeks of the consent date due to an unregulated systemic disease.
5. Severe MGD patient
6. Ophthalmic surgery (including Lasik/Lasek) and trauma in eyes within the last three months
7. Wearing contact lenses during a clinical trial period
8. Planning an eye surgery (including Lasik/Lasek) during the clinical trial period
9. Hypersensitivity to the clinical trial drug
10. Active or suspected eye infections
11. Pregnant or breastfeeding, or women planning to become pregnant
12. Participation in other clinical trials within three months
13. Any person who is deemed unfit for clinical trial by a investigator

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Cornea staining score (NEI scale) | 12 weeks
  The cornea staining score(NEI scale) is a grading scale for the corneal surface after fluorescein staining to help measure the efficacy of dry eye treatment. A standardized grading system of 0 to 3 is used for each of the five areas on each cornea. Grade 0 is specified when no staining is present, and the maximum score is 15.

SECONDARY OUTCOMES:
Ratio of patients who have improvement, deterioration, and no-change of cornea staining scores(NEI scale) | 4 weeks, 8 weeks, 12 weeks
  Cornea staining scores (NEI scale) (Improvement: decrease by more than one point / Deterioration : increase by more than one point / No change: no change in score)
Conjunctival staining scores (NEI scale) | 4 weeks, 8 weeks, 12 weeks
  The conjunctival staining score(NEI scale) is a grading scale for the conjunctival surface after fluorescein staining to help measure the efficacy of dry eye treatment. A standardized grading system of 0 to 3 is used for each of the six areas on each conjunctiva. Grade 0 is specified when no staining is present, and the maximum score is 18.
Tear Break-Up Time (TBUT) | 4 weeks, 8 weeks, 12 weeks
  Tear Break-Up Time(TBUT) is a clinical test used to evaluate the dry eye disease after the fluorescein is instilled into the patient's tear film.
SANDE(Symptom Assessment in Dry Eye) score | 4 weeks, 8 weeks, 12 weeks
  SANDE (Symptom Assessment in Dry Eye)is a short questionnaire that quantifies both severity and frequency of dry eye symptoms
Tear Meniscometry score | 4 weeks, 8 weeks, 12 weeks
  A simple method of quantification of the volume of tear meniscus in the diagnosis of the dry eye syndromes.
ODS (Ocular Discomfort Scale) | 4 weeks, 8 weeks, 12 weeks
  A simple questionnaire to evaluation the dry eye symptom of stinging, irritation, itching, and blurred vision.(0 to 10 points)
Patient Reported Outcome (PRO) | 12 weeks
  A short questionnaire to evaluation the improvement of dry eye symptom by a patient.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Yul Seo, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No